CLINICAL TRIAL: NCT04691830
Title: Adaptation of a Rehabilitation Program for Prosody and Its Application on Egyptian Hearing Impaired Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Magdy Ibrahim (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Sara Magdy Ibrahim, Demonstrator of phoniatrics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0105832
Record Dates: First submitted 2020-12-28; First posted 2020-12-31 (Actual); Last update posted 2020-12-31 (Actual); Status verified 2020-12

CONDITIONS: Hearing Impaired Children
Keywords: Hearing impairment; Prosody; Speech rehabilitation; Cochlear implant
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: a comparative intervention study comparing the effect of prosodic rehabilitation in addition to the traditional language and auditory training on prosodic skills of hearing impaired children in comparison to traditional language and auditory rehabilitation alone.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group IA (Experimental): Preschool cases group who received the proposed "prosody treatment program" in addition to the traditional auditory and language rehabilitation therapy.
  Interventions: Behavioral: Prosody treatment program; Behavioral: Traditional auditory and language rehabilitation
- group IB (Active Comparator): preschool control group who received the traditional auditory and language rehabilitation therapy without the prosody rehabilitation program. This was considered the preschool age control group.
  Interventions: Behavioral: Traditional auditory and language rehabilitation
- group IIA (Experimental): School age cases group who received the proposed "prosody treatment program" in addition to the traditional auditory and language rehabilitation therapy.
  Interventions: Behavioral: Prosody treatment program; Behavioral: Traditional auditory and language rehabilitation
- group IIB (Active Comparator): School age control group who received the traditional auditory and language rehabilitation therapy without the prosody rehabilitation program. This was considered the school age control group.
  Interventions: Behavioral: Traditional auditory and language rehabilitation

INTERVENTIONS:
Behavioral: Prosody treatment program — The "prosody treatment program" is an evidence-based practice targeting receptive and expressive prosodic skills in addition to speech production, intelligibility, pragmatics and phonology. The program incorporates the principles of validated prosodic rehabilitation strategies such as Dynamic Temporal and Tactile Cueing (DTTC), Melodic Intonation Therapy, Lee Silverman Voice Treatment in addition to expert professional practice.
  The program was applied using a systematic approach of providing cues to help accelerate the child's learning of the prosodic skills targeted in the program. The program is divided into two sections according to the age into preschool section and school age section.
  Arms: group IA; group IIA
Behavioral: Traditional auditory and language rehabilitation — Auditory rehabilitation therapy included activities targeting auditory skills: sound detection, discrimination, identification and auditory comprehension. Language rehabilitation targeted improving semantics, syntax, pragmatics and phonology.

SUMMARY:
Prosody is the melody and rhythm of speech, it is used to refer to the supra segmental aspects of speech including pitch, loudness and duration. Variations in these features achieve different prosodic functions and are perceived by the listener as meaningful changes. The role of prosody in language acquisition and effective communication is documented in research. Nevertheless, prosodic intervention in children with hearing impairment received less attention compared to other speech and language areas.

The aim of this study is to adapt the "prosody treatment program", an evidence based rehabilitation program, and to detect the efficacy of its activities in improving the prosodic skills of Egyptian hearing impaired children.

The "prosody treatment program" is an evidence-based practice targeting receptive and expressive prosodic skills in addition to speech production, intelligibility, pragmatics and phonology. The program is applied using a systematic approach of providing cues following the principles adapted from dynamic temporal and tactile cueing (DTTC) for speech motor learning to help accelerate the child's learning of the prosodic skills targeted in this program. The program was translated to Arabic and adapted to be suitable for the Egyptian children.

DETAILED DESCRIPTION:
Prosody has an important role in several areas of communicative functions including : grammatical, pragmatic, affective and/or indexical functions. Prosodic abnormalities extend across a wide range of communication disorders. Intact functioning auditory system has a fundamental role in language acquisition and development. Children receive the speech of others as a source of linguistic input which is considered their target and they gradually modify their productions using their own auditory feedback to reach the target utterance.

Hearing impairment early in life deprives the child of the source of their linguistic input affecting various aspects of speech and language development. Speech production of the hearing impaired is characterized by various segmental and suprasegmental errors.

Case studies show that interventions targeting prosody can modify prosody in young children with speech and language impairments. Multiple problems of prosody , language, speech and voice are found in individuals with prosodic impairments ,therefore it is challenging to develop treatment protocols addressing prosody .There are only few published interventions targeting prosody .

Due to lack of well structured comprehensive Arabic programs targeting prosody , this work was dedicated towards adaptation of "prosody treatment program" a remediation program targeting receptive and expressive prosodic skills and its application on hearing impaired children .The proposed program targets two levels: preschool and school aged children.

The aim of this work was to adapt the "prosody treatment program" program and apply its activities in cases of hearing impairment to detect its efficacy in improvement of prosodic skills in Egyptian hearing impaired children fitted with hearing aids or cochlear implant devices.

This study was conducted on 55 children with hearing impairment attending the Unit of Phoniatrics , in the outpatient clinic of Alexandria Main University hospital. Sample size was calculated using two proportions power analysis in NCSS and PASS program a minimum sample size required to detect the efficacy of the "prosody treatment program" in improvement of prosodic skills of Egyptian hearing impaired children and to detect a difference of 0.5 that achieve 80% power with a target significance level at 5%.

The proposed program is based on " prosody treatment program", a program targeting receptive and expressive prosodic skills. It includes activities targeting loudness , word stress ,syllable stress ,pitch ,question inflections ,emotions ,sarcasm ,rhythm ,chunking, and speaking rate . The program was adapted in order to be appropriate to the Arabic language and to the Egyptian children. The program was applied using a systematic approach of providing cues to help accelerate the child's learning of the prosodic skills targeted in the program. Cues are adapted from the Dynamic Temporal and Tactile Cueing (DTTC) for Speech Motor Learning hierarchy. It aims at improving motor planning, and programming speech processing as speech and language acquisition progresses.

The program is divided into two sections according to the age into preschool section and school age section.

A pilot study was conducted on 8 cases with hearing impairment attending the phoniatrics unit to check the suitability of the rehabilitation program and modify the needed items.

All subjects met the specified inclusion and exclusion criteria and were assessed by the specified protocol of assessment to evaluate prosodic skills, language skills and cognitive abilities before and after intervention.

Data were analyzed using IBM SPSS software package version 20.0. (Armonk, NY: IBM Corp). Qualitative data were described using number and percent. Chi square test was used for comparison of qualitative variables in two groups, Fisher exact test was used to compare qualitative variables when 50% of cell value was less than 5. McNemar test was used to compare nominal variables before and after intervention. The Kolmogorov-Smirnov test was used to verify the normality of distribution. Quantitative data were described using mean, standard deviation and IQR. Test of significance used included different tests. t test to compare between different means. Mann Whitney U test to compare non normally distributed quantitative variables in two different groups. Paired t test for comparison of normally distributed variables in matched pairs. Wilcoxon signed rank test for pre-post comparison in non-normally distributed quantitative variables. Kappa coefficient was used to assess level of agreement between two raters. Significance of the obtained results was judged at the 5% level.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impaired children of both sexes, in the preschool age (from 3 to 6 years), and school age (6 to 18 years).
* Children using auditory verbal communication.
* Children with moderately severe or severe up to profound sensorineural hearing loss in unaided conditions, fitted with hearing aids or cochlear implant devices with good benefit (aided hearing threshold less than 40 dB across all frequencies).

Exclusion Criteria:

* Children with intellectual disability.
* Children with brain damage.
* Children with additional sensory deprivation (impaired vision).
* Psychiatric problems (example; ASD).
* Motor speech disorders (example: apraxia, dysarthria).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2020-02-16 (Actual); Study Completion 2020-02-16 (Actual)

PRIMARY OUTCOMES:
change in prosodic skill assessment protocol subjective measures | baseline and 3 months
  a quantitative test that evaluates ten prosodic skills, each skill is given a subjective score from 0 to 4 (4 is the best score) with a total score of 40.
change in prosodic skill assessment protocol mean frequency measures | baseline and 3 months
  a quantitative tool that evaluates mean frequency value of recorded utterances in hertz
change in prosodic skill assessment protocol mean duration measures | baseline and 3 months
  a quantitative tool that evaluates mean duration of recorded utterances in msec
change in prosodic skill assessment protocol mean energy measures | baseline and 3 months
  a quantitative tool that evaluates mean energy of recorded utterances in dB
Change in Arabic prosodic assessment tool subjective ratings | baseline and 3 months
  a qualitative tool that rates prosodic skills of recorded utterances as either (A) Appropriate or (I) Inappropriate
Change in Arabic prosodic assessment tool frequency measures | baseline and 3 months
  a quantitative tool that evaluates frequency values of recorded utterances in hertz
Change in Arabic prosodic assessment tool duration measures | baseline and 3 months
  a quantitative tool that evaluates duration of recorded utterances in msec
Change in Arabic prosodic assessment tool energy measures | baseline and 3 months
  a quantitative tool that evaluates energy of recorded utterances in dB

SECONDARY OUTCOMES:
change in Arabic language test scores | baseline and 3 months
  a quantitative too that evaluates language skills, raw scores are converted into language age equivalent scores
change in values of Stanford Binet scale | baseline and 3 months
  a quantitative tool that evaluates intelligence quotient

CONTACTS AND LOCATIONS:
Overall Officials: Ossama A Sobhy, PhD, Principal Investigator — Alexandria University; Rania M Abdou, PhD, Study Chair — Alexandria University; Nesrine H Hammouda, PhD, Study Director — Alexandria University; Sara M Ibrahim, Master's, Study Director — Alexandria University
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sobhy OA, Abdou RM, Ibrahim SM, Hamouda NH. Effects of Prosody Rehabilitation on Acoustic Analysis of Prosodic Features in Hearing-Impaired Children: A Randomized Controlled Trial. Folia Phoniatr Logop. 2022;74(1):29-45. doi: 10.1159/000516979. Epub 2021 Jul 21. PMID 34289481